CLINICAL TRIAL: NCT06253689
Title: Impact of Defecation Posture on Ease of First Bowel Movement Following Posterior Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-087
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Constipation; Pelvic Organ Prolapse Vaginal Surgery; Defecation Function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Defecation Posture Modification Device (Experimental)
  Interventions: Device: Defecation Posture Modification Device
- Control (No Intervention)

INTERVENTIONS:
Device: Defecation Posture Modification Device — Patients assigned to the experimental arm will be asked to use the defecation posture modification device to aid with bowel movements during the postoperative period.
  Other Names: Squatty potty
  Arms: Defecation Posture Modification Device

SUMMARY:
This study will determine if defecation posture, when using a defecation posture modification device (DPMD), improves ease with first bowel movement following pelvic reconstructive surgery, specifically posterior repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery by one of the sub investigators including a posterior compartment repair

Exclusion Criteria:

* Anyone currently using a defecation posture modification device
* Unwillingness or unable to participate in the study
* Presence of ileostomy/colostomy
* Wheelchair bound
* Device may pose fall or safety hazard risk to patient
* Patients weighing over 250 lbs, as per device manufacturer guidelines
* Inability to understand English
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Straining with first postoperative bowel movement | 1 week
  patients will keep 7 day log of each postoperative bowel movement within the first week of surgery, they will assess with an 11 point numeric rating scale their level of strain with bowel movement, the scale starts at 0 indicating no straining and 10 indicating maximal straining/effort. I high score of 10 means a worse outcome. The scale title is "straining with bowel movement".

SECONDARY OUTCOMES:
postoperative stool consistency | 1 week
  7 day bowel movement diary using bristol stool scale to describe stool consistency. The Bristol Stool scale is a validated scale to describe each type stool consistency. The scale is from Type 1 - Type 7. Type 1 is separate hard lumps of stool and ranges up to Type 7 which is watery and entirely liquid stool. In this scale the two ends (high and low) are concerned worse outcomes, the middle of the scale - Type 4 is the ideal outcome.
Time to first bowel movement | 1 week
  7 day log for patients to track bowel movements within 1st week of surgery
pain with postoperative bowel movements | 1 week
  7 day log where patients input each bowel movement for the first week postoperative, 11 point numeric scale for tracking pain. The scale is a pain rating scale with 0 indicating no pain with bowel movements and 10 indicating worst possible pain with bowel movements. The title of the scale is "Pain with bowel movements". The worse outcome is a 10 and the best outcome is a zero.
Postoperative use of laxatives and pain medication | 1 week
  patients will keep 7 day log of daily usage of standard postoperative pain medication and laxative use
Satisfaction with device and ease of use | 1 month
  patients will receive a questionnaire with questions regarding their satisfaction with the device and ease of use. When asked about satisfaction of the device, patients will be given an 11 point numeric scale assessing satisfaction. The number 0 will indicate not satisfied and 10 will indicate very satisfied with use of the device. The title of the scale is "satisfaction with device". The Best outcome is a 10 and the worst outcome is a 0.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cincinnati Urogynecology Associates, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No